CLINICAL TRIAL: NCT00327522
Title: An Open, Phase I/II Study to Evaluate the Safety, Reactogenicity and Immunogenicity of GSK Biologicals' 11PCV Vaccine Given as a 2-Dose Vaccination in Adults Aged 18-40 Years Old.
Brief Title: Safety and Immune Response Study of an Investigational Pneumococcal Vaccine.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 106962; NCT00309153 (obsolete NCT alias)
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Prophylactic Pneumococcal Diseases
MeSH Terms: interventions — Pneumococcal Vaccines

INTERVENTIONS:
Biological: pneumococcal vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of two doses of GSK Biologicals' 11 PCV vaccine when given to healthy subjects aged 18 to 40 years .

DETAILED DESCRIPTION:
The study is open and subjects will receive two vaccine doses of GSK Biologicals' 11 PCV vaccine. Five blood samples will be taken: prior to and one month after each vaccine dose, and 2 weeks after dose 2.

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female between 18 and 40 years of age
* 23-valent pneumococcal polysaccharide vaccine naive adults.

Exclusion Criteria:

* Previous vaccination against Streptococcus pneumoniae.
* History of pneumonia within 3 years prior to the first vaccination
* Any confirmed or suspected immunosuppressive or immunodeficient condition
* All malignancies (excluding non-melanic skin cancer) and lymphoproliferative disorders diagnosed or treated actively during the past 5 years.
* Subjects with documented anaemia or iron-deficiency (Hemoglobin level more than 10% below lower limit of normal)
* History of administration of an experimental/licensed vaccine containing similar adjuvants.
* History of chronic alcohol consumption and/or drug abuse.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2006-06

PRIMARY OUTCOMES:
Occurrence of solicited local & general symptoms (Day 0-7) and unsolicited symptoms (Day 0-30) after vaccination. Occurrence of serious adverse events during the entire study;
Frequencies of IgG PS-specific plasma cells (by B-cell ELISPOT) for 11 serotypes (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, 23F) prior to & 1 month post dose 1, 2 weeks & 1 month post dose 2

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium